CLINICAL TRIAL: NCT03763799
Title: Impact of a Strategy Based on the Unyvero® Testing System on Appropriate Antimicrobial Treatment in Patients With Suspected Aspiration Pneumonia Requiring Mechanical Ventilation : a Randomized Controlled Unblinded Trial
Brief Title: Early Stop(Ruling) of the Antibiotic Treatment During Pneumopathies d' Inhalation
Acronym: APAPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018_40; 2018-A02219-46 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-12-03; First posted 2018-12-04 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Aspiration Pneumonia
Keywords: Aspiration pneumonia; Invasive ventilation; PCR; Antibiotics; Tracheal aspirate
MeSH Terms: conditions — Pneumonia, Aspiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multiplex PCR strategy (Experimental): FilmArray® Pneumonia Panel plus
  Interventions: Procedure: PCR-based microbiological diagnosis strategy
- standard strategy (Active Comparator)
  Interventions: Procedure: Standard microbiological diagnosis strategy

INTERVENTIONS:
Procedure: PCR-based microbiological diagnosis strategy — A multiplex PCR-based testing, will be used in addition to standard microbiological culture of the tracheal aspirate to diagnose bacterial pneumonia after inhalation
  Arms: multiplex PCR strategy
Procedure: Standard microbiological diagnosis strategy — Standard strategy will be based on with standard microbiological culture of the tracheal aspirate to diagnose bacterial pneumonia after inhalation
  Arms: standard strategy

SUMMARY:
The two most common consequences resulting from aspiration are chemical pneumonitis and bacterial aspiration pneumonia. Both entities present with comparable clinical signs and symptoms. In the absence of a reliable clinical or biological marker to differentiate between these two conditions, most patients with suspected aspiration are treated empirically with antibiotics. De-escalation of initial antibiotic treatment is encouraged based on the results of microbiological results, usually performed before starting antimicrobial treatment. However, in most hospitals, 48-72h are required to obtain the results of microbiological cultures, and to de-escalate empirical large spectrum antibiotic treatment.

The use of the Unyvero®, a multiplex PCR-based testing system, for detection of respiratory bacterial pathogens would allow decreasing the percentage of patients with aspiration syndrome who will receive unappropriated antibiotic treatment at Day 3.

ELIGIBILITY:
Inclusion Criteria:

* presence of risk factors for aspiration :
* known or likely swallowing dysfunction,
* altered consciousness,
* cardiac arrest,
* difficult intubation
* witnessed aspiration
* symptoms and signs suggestive of lower respiratory tract pathology
* temperature ≥38.5°C or <36°C
* leukocyte count ≥10 000/µL or <1500/µL
* purulent sputum or tracheal aspirate.
* new radiographic infiltrate on chest X-ray
* tracheal intubation and mechanical ventilation since less than 48 hours

Exclusion Criteria:

* pregnant women
* refuse to participate to the study
* no informed consent
* documented bacteremia
* septic shock
* severe immunosuppression: leukocytes<1000/L or neutrophils<500/L, chemotherapy during the last 3 months, organ transplant with chronic immunosuppressors use, HIV (CD4<50), and chronic corticosteroid use (>0.5 mg/kg day for at least one month during the last three months).
* moribund patients (SAPS II >90).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
The percentage of patients who will benefit from an early stop of the probabilist antibiotic treatment | 48 hours after antibiotic treatment initiation

SECONDARY OUTCOMES:
the percentage of patients who will receive appropriate antibiotic treatment. | at Day 28 and Day 90 after antibiotic treatment initiation
the percentage of patients who will receive targeted antibiotic treatment. | at Day 28 and Day 90 after antibiotic treatment initiation
mechanical ventilation free days. | at Day 28 and Day 90 after antibiotic treatment initiation
length of ICU stay. | up to Day 90
ICU mortality. | up to Day 90
antibiotic free days. | up to Day 90
percentage of patients with colonization or infection related to multidrug-resistant bacteria (MDR) | at Day 28 and Day 90 after antibiotic treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Saadalla NSEIR, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (2):
- France (2):
  - Chu Amiens Picardie, Amiens
  - Hôpital Roger Salengro, CHU, Lille